CLINICAL TRIAL: NCT01917604
Title: Oral Health Related Quality of Life and Clinical Outcomes in Patients Undergoing Canine Disimpaction- A Randomized Control Trial.
Brief Title: Oral Health Related Quality of Life and Clinical Outcomes in Patients Undergoing Canine Disimpaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jamia Millia Islamia (Other)
Collaborators: Council of Scientific and Industrial Research, India (Other Government)
Responsible Party: Principal Investigator, DR.PANCHALI BATRA, Professor, Department of Orthodontics, Jamia Millia Islamia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: imc25
Record Dates: First submitted 2013-08-01; First posted 2013-08-06 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Tooth, Impacted
Keywords: Open versus Closed surgical technique; Palatally impacted maxillary canine; Orthodontic disimpaction; Oral health related Quality of life
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open exposure and control (Experimental): ● surgically uncover the canine tooth and bone removal exposing the largest diameter of the ectopic canine crown make a window in the palatal soft tissue and bond bracket after 10 days
  Interventions: Procedure: open exposure
- closed exposure and control (Experimental): raising a flap in the area of impacted canine,bonding an attachment and resuturing the flap
  Interventions: Procedure: closed exposure

INTERVENTIONS:
Procedure: open exposure — the open surgical methods of exposing the canine is compared with control
  Arms: open exposure and control
Procedure: closed exposure — closed exposure is compared with control
  Arms: closed exposure and control

SUMMARY:
To test the null hypothesis that there are no differences in the OHRQOL and clinical outcomes in patients undergoing palatal canine disimpaction using either open or closed surgical method.

DETAILED DESCRIPTION:
The study design will be a unicentric, randomized controlled clinical trial involving 2 parallel groups. The protocol has been approved by local ethics committee of Jamia Millia Islamia and all participants will be provided with an informed consent agreement. The settings will be the orthodontic department of a dental teaching hospital (Faculty of Dentistry, Jamia Millia Islamia). Participants for the trial will be identified from treatment waiting lists and new patient clinics.

Proper randomization procedures and reporting include the following steps.

1. Generation of the random allocation sequence, including details of any restrictions.
2. Allocation concealment.
3. Implementation of the random allocation sequence:

information on who generated the allocation sequence, who enrolled the participants, and who assigned them to their groups.

OPEN SURGICAL EXPOSURE

* Surgically uncover the canine tooth followed by bone removal exposing the largest diameter of the ectopic canine crown. The edges need to be substantially trimmed back and dental follicle removed to prevent reclosure of the very thick palatal mucosa.
* Surgical excision of the palatal mucosa-standardized using a preformed wire template.
* Coe-pack surgical dressing (GC America Inc, Alsip, IL) will be left in place.
* The patient will be reviewed 10 days later and the surgical pack removed and the bracket bonded and force application started once the tooth has erupted sufficiently for an orthodontic attachment to be glued onto its surface, orthodontic brace treatment is commenced to bring the tooth into line.

CLOSED SURGICAL EXPOSURE

• Surgically uncover the canine tooth and Surgical bone removal exposing the largest diameter of the ectopic canine crown.

* An multipurpose attachment with ligature wire and e chain will be bonded to the palatal or buccal surface of the ectopic canine crown (whichever was the most accessible).
* An orthodontic attachment (button) with ligature wire and bracket with closed coil spring will be bonded to the palatal or buccal surface of the ectopic canine crown (whichever was the most accessible).

Outcome Assessment:

The following outcomes will be measured before, during and post orthodontic treatment:

Primary Outcome Measures:

1. Oral health based Quality of life of patients undergoing canine disimpaction will be accessed by questionnaire pre-treatment and post treatment (one month after debond) -(Annexure 1 - page 1,2)
2. Oral health based Quality of life of patients undergoing canine disimpaction will be accessed by questionnaire 24 hrs and 10 days after surgical caniine exposure (Annexure 1 - page 3,4).
3. Measurement of clinical outcomes 3 months post debond (details mentioned in Annexure 2).
4. Maxillary Canine Aesthetic Index (one month after debond) - Annexure 3

ELIGIBILITY:
Inclusion Criteria:Patients with palatally ectopic maxillary canines who required surgical exposure and orthodontic alignment

* Age 13-25 years Minimal orthodontic problems other than the ectopic canine
* Good oral hygiene and motivated to wear fixed appliances for at least 2 years

Exclusion Criteria:

Compromising medical conditions (patients requiring antibiotic prophylaxis to prevent infective endocarditis)

* Periodontal disease (bleeding on probing, pocket probing depths _3 mm and decreased bone levels as diagnosed from baseline panoramic imaging)
* Cases in which the canine is to be brought into the position of the lateral incisor.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Oral health based Quality of life (Annexure 1; page 1 and page 2) | pre-treatment and 1 month post treatment (average duration of treatment 18 months )
  to evaluate change in Oral health based Quality of life of patients undergoing canine disimpaction will be accessed by questionnaire and compared for both groups
Post- surgical Oral health based Quality of life (24 hours after surgical exposure) (Annexure 1; page 3) | 24 hours after surgical exposure
  Post- surgical Oral health based Quality of life of patients undergoing canine disimpaction will be accessed by questionnaire and compared for both open and closed groups
Post- surgical Oral health based Quality of life (10th day after surgical exposure)(Annexure 1; page 4) | 10th day after surgical exposure
  Post- surgical Oral health based Quality of life of patients undergoing canine disimpaction will be accessed by questionnaire and compared for both open and closed groups
Clinical outcomes - periodontal (Annexure 1; page 5) | Three month post debond
  Periodontal outcomes of disimpacted canines accessed clinically and compared for both open and closed groups; contralateral canine of maxillary arch will be control group.
Maxillary canine aesthetic index (Annexure 1; page 7) | one month after debond
  comparision to control side with experimental side of both the groups

CONTACTS AND LOCATIONS:
Overall Officials: panchali batra, m.d.s., Principal Investigator — Jamia Millia Islamia
Locations (1):
- Jamia Millia Islamia, Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Parkin NA, Deery C, Smith AM, Tinsley D, Sandler J, Benson PE. No difference in surgical outcomes between open and closed exposure of palatally displaced maxillary canines. J Oral Maxillofac Surg. 2012 Sep;70(9):2026-34. doi: 10.1016/j.joms.2012.02.028. Epub 2012 Jun 6. PMID 22677328

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT01917604/Prot_ICF_000.pdf